CLINICAL TRIAL: NCT05204316
Title: NLP Headache Speech (NLPH-SPEECH): a Cross-sectional Study on Natural Language Processing Analysing Spoken Monologues by Headache Patients
Acronym: NLPH SPEECH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BC-10619
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Headache Disorders
MeSH Terms: conditions — Headache Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): Participants will provide spoken narratives on their headache disorder
  Interventions: Other: Digital Analysis of Speech

INTERVENTIONS:
Other: Digital Analysis of Speech — Recordings will be transcribed manually to written digital text formats, on which NLP tools such as tokenisation and lexical analysis will be performed.

SUMMARY:
The research collects spoken descriptions of headache disorders by participants with headache disorders. The speech recordings are analyzed by natural language processing (NLP) tools to analyse linguistic properties of the texts and to obtain insight into the potential of NLP machine learning models for the recognition of headache syndromes of the participants.

ELIGIBILITY:
Inclusion Criteria:

* is a patient of the tertiary headache clinic at Ghent University Hospital
* is 18 years or older
* has Dutch as native speaking language

Exclusion Criteria:

* has difficulties in producing spoken language
* has limited or no knowledge of Dutch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Linguistic analysis of texts | through study completion, an average of 1 year
  Descriptive linguistic analysis of lexical choices, sentence formation and thematic content within the texts

SECONDARY OUTCOMES:
Machine learning modelling for classification of headache disorders | through study completion, an average of 1 year
  To investigate the potential and learn insights of machine learning modelling to classify headache disorders based on the descriptions by participants
Machine learning modelling for estimation of headache impact scores | through study completion, an average of 1 year
  To investigate the potential and learn insights of machine learning modelling to estimate headache impact scores from different validated questionnaires investigating burden of disease and quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Gent - Dienst Neurologie, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No
Strict secured storage of IPD on Ghent University Hospital servers.